CLINICAL TRIAL: NCT00893685
Title: Elderly Friendly Alarm Handling and Monitoring (DREAMING)
Brief Title: Randomized Controlled Trial of Home Telemonitoring for Elderly People
Acronym: Dreaming
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Health Information Management, Belgium (Other)
Responsible Party: Marco D'Angelantonio, Health Information Management Sa, Belgium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: European Commission; European Commission; ICT support policy program; Contract Number 225023
Record Dates: First submitted 2009-04-22; First posted 2009-05-06 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus; Chronic Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Telemedicine
MeSH Terms: conditions — Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home telemonitoring (Experimental)
  Interventions: Device: Wireless monitors for disease specific clinical parameters.
- Usual care (control group) (No Intervention)

INTERVENTIONS:
Device: Wireless monitors for disease specific clinical parameters. — Homes of participants will be equipped with wireless monitors for blood pressure, blood oxygen, blood glucose, peak expiratory flow, electrocardiogram, body weight. All vital parameters are monitored on a continuous, at least daily basis and obtained values are transmitted to a monitoring centre. Abnormal values are classified for their health risk and health alarms and/or intervention of health professionals is triggered.
  Arms: Home telemonitoring

SUMMARY:
The DREAMING clinical trial is part of the DREAMING project, which has the objective to demonstrate that the DREAMING platform consisting of integrated health monitoring, alarm handling and videoconferencing services produces clinical benefits to its users and economic benefits to the health authorities. The study evaluates the long-term (30 months) effect of continuous use of the DREAMING subsystems and is testing the hypothesis that such use is superior to usual care alone in reducing the deterioration of health related quality of life that is associated to age and chronic disease. It also tests the hypothesis that the DREAMING environment is superior to usual care in delaying the transfer to nursing or elderly homes and in reducing the incidence and duration of hospitalisation episodes. The trial will also evaluate the cost-effectiveness of the DREAMING platform. Outcomes are assessed in six different health care systems (Denmark, Estonia, Germany, Italy, Spain and Sweden) and will represent a basis for the adoption of DREAMING services by the respective health authorities.

DETAILED DESCRIPTION:
Homes of participants are equipped with environmental sensors, motion detection, and with wireless sensors for blood pressure, blood glucose, body weight, blood oxygen saturation, peak expiratory flow and electrocardiogram. Disease related parameters are monitored at least daily and the measured values are transmitted to a central monitoring unit. In case of abnormal values, health alarms are generated and transmitted to the local health authorities to trigger eventual intervention by the physicians and nurses who normally follow the participants. Participants and health professionals can stay in contact via an easy to use, home television based videoconferencing system. Participants are also equipped with a a personal alarm and GPS-enhanced localisation system.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Diagnosis of chronic heart failure
* Diagnosis of diabetes mellitus
* Diagnosis of chronic obstructive pulmonary disease

Only in the case that the number of recruited participants is not sufficient, inclusion criteria can be extended to one or more of the following conditions:

* History of myocardial infarction
* History of stroke (brain ischemia or hemorrhage)
* History of falls within the last two years
* Hospitalization during the last two years (for every reason)

Exclusion Criteria:

* Not willing to participate (e.g non signing informed consent)
* Inability to use the DREAMING equipment
* Significant impairment of language comprehension or expression (aphasia)
* Diagnosis of dementia
* Completely dependent on others for the activities of daily living
* Living without access to ISDN or DSL service

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life as assessed by the SF-36 questionnaire, at the beginning, at midterm and at the end of the trial period | 0, 15, 30 months

SECONDARY OUTCOMES:
Time to permanent transfer to elderly homes | Measured at month 30
Total and average length of stay in hospital | Measured at month 30
Number of consultations with general practitioners | Measured at month 30
Number of consultations with medical specialists | Measured at month 30
Number of home visits by nurses | Measured at month 30
Number of ambulance transports | Measured at month 30
Number of accesses to emergency rooms | Measured at month 30
Number of falls | Measured at month 30
Number of femur fractures | Measured at month 30
HbA1c change over time (only for participants with a diagnosis of diabetes) | Measured at month 30
Survival | Measured at month 30
Depression as measured by HADS | Measured at months 0, 15 and 30
Number of hospitalisations | Measured at month 30
Number of permanent transfers to elderly homes | Measured at month 30

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard W Prior, M.D., Study Director — Health Information Management, Brussels, Belgium; Helmut Prior, Prof. Dr., Principal Investigator — Institute for Experimental Psychology, University of Düsseldorf, Germany (H.Prior is head of the data monitoring committee)
Locations (6):
- Langeland Municipality, Langeland, Denmark
- East Tallin Central Hospital, Tallinn, Estonia
- Pflegwerk Berlin, Mediplus, Berlin, Germany
- Azienda per i Servizi Sanitari ASS N.1, Trieste, Italy
- Servicio Aragones de Salud, Barbastro, Spain
- GP Surgery, Heby, Sweden